CLINICAL TRIAL: NCT06507904
Title: A Phase 1, Randomized, Crossover Design Study to Assess Palatability of Osivelotor (PF-07940367) Pediatric Formulations With Dosing Vehicle (Part 1) and Randomized, Single-Dose, Parallel Design Study to Estimate Relative Bioavailability of Osivelotor Pediatric Formulation With Dosing Vehicle and With Water Compared to Clinical Tablet Formulation, and Effect of Food and/or Acid-Reducing Agent On Bioavailability In Healthy Adult Participants (Part 2)
Brief Title: A Study to Learn How Different Preparations of Osivelotor Taste and Enter the Blood With Food or Liquids or With an Antacid in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: C5351009; 2024-511410-20-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: palatability; bioavailability
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 Sequence 1 - Palatability (Experimental): Participants will receive 4 preparations (Treatments A, B, C, D) of osivelotor pellet/granules at least 2 hours apart on Day 1 which they will put in their mouth and then spit it out.
  Interventions: Drug: Osivelotor
- Part 1 Sequence 2 - Palatability (Experimental): Participants will receive 4 preparations (Treatments B, C, D, A) of osivelotor pellet/granules at least 2 hours apart on Day 1 which they will put in their mouth and then spit it out.
  Interventions: Drug: Osivelotor
- Part 1 Sequence 3 - Palatability (Experimental): Participants will receive 4 preparations (Treatments C, D, A, B) of osivelotor pellet/granules at least 2 hours apart on Day 1 which they will put in their mouth and then spit it out.
  Interventions: Drug: Osivelotor
- Part 1 Sequence 4 - Palatability (Experimental): Participants will receive 4 preparations (Treatments D, A, B, C) of osivelotor pellet/granules at least 2 hours apart on Day 1 which they will put in their mouth and then spit it out.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment E (Experimental): Participants will receive 1 preparation (Treatment E) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment F (Experimental): Participants will receive 1 preparation (Treatment F) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow. They might have a dose on Day 7 which they will put in their mouth and then spit it out; afterwards they will complete the taste questionnaire.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment G (Experimental): Participants will receive 1 preparation (Treatment G) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment H (Experimental): Participants will receive famotidine and afterwards preparation (Treatment H) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow.
  Interventions: Drug: Osivelotor; Other: Famotidine
- Part 2 Pharmacokinetics - Treatment I (Experimental): Participants will receive 1 preparation (Treatment I) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment J (Experimental): Participants will receive 1 preparation (Treatment J) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow. They might have a dose on Day 7 which they will put in their mouth and then spit it out; afterwards they will complete the taste questionnaire.
  Interventions: Drug: Osivelotor
- Part 2 Pharmacokinetics - Treatment K (Experimental): Participants will receive 1 preparation (Treatment K) of osivelotor pellet/granules on Day 1 which they will put in their mouth and swallow.
  Interventions: Drug: Osivelotor

INTERVENTIONS:
Drug: Osivelotor — A medicine to treat sickle cell disease.
  Other Names: PF-07940367
Other: Famotidine — Famotidine is a marketed medicine which decreases the amount of acid made in the stomach and is used to prevent and treat heartburn.
  Arms: Part 2 Pharmacokinetics - Treatment H

SUMMARY:
A study to learn how different preparations of Osivelotor taste and enter the blood with food or liquids, or with an antacid in healthy adults.

DETAILED DESCRIPTION:
This study has two parts: Part 1 and Part 2. The purpose of Part 1 of this study is to learn how different preparations of the study medicine called osivelotor (PF-07940367) taste. The purpose of Part 2 of this study is to learn how the study medicine is taken up into the blood when mixed with:

* soft foods or liquids given on an empty stomach or
* with an acid-reducing agent in healthy adults.

This study is seeking participants who are:

* healthy females and males of 18 to 65 years of age.
* have a body mass index of 16 to 32 kilogram per meter squared.
* have a total body weight of more than 50 kilograms (110 pounds).

Participants in Part 1 of the study will receive the study medicine 4 times with at least 2-hour interval on day one. This study medicine will not be swallowed but will be placed in the mouth and spat out. The participants will then complete a short questionnaire 4 times over 20 minutes. All study medicines will be given in the study clinic.

Participants in Part 2 of the study will receive the study medicine up to 2 times. The first dose of the study medicine will be swallowed. The second dose the study medicine (if given) will not be swallowed but will be placed in the mouth and spat out for the taste questionnaire as above. All study medicines will be given in the study clinic.

In Part 1, participants will be involved in this study for up to 2 months. During this time, there will be a two-day stay in the study clinic. After leaving the clinic, study team will also call participants once over the phone. Woman who could become pregnant may need to visit the study clinic instead of receiving a phone call.

In Part 2, participants will be involved in this study for up to 4 months. During this time, there will be a seven-day stay in the study clinic. After leaving the clinic, the study team will also call participants 3 times over the phone. Woman who could become pregnant may need to visit the study clinic instead of receiving a phone calls.

In both parts blood and urine tests will be done, and blood pressures and heart traces taken. Also, contraception requirements will need to be followed to prevent pregnancy during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years (or the minimum age of consent in accordance with local regulations if >18 years) to 65 years (inclusive) at screening who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination (PE), including blood pressure (BP) and pulse rate (PR) measurement, 12-lead ECG (electrocardiogram) and clinical laboratory tests.
* Body mass index (BMI) of ≥16 to ≤32 kg/m2; Body weight ≥50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Use of prescription or nonprescription drug, dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer), with the exception of moderate or strong cytochrome P450 (CYP)3A inducers or inhibitors which are prohibited within 14 days plus 5 half-lives, prior to the first dose of study intervention.
* Current use of any prohibited concomitant medication(s) or participant unwilling/able to use a permitted concomitant medication(s).
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* For females, pregnancy, as indicated by a positive serum pregnancy test (serum) at screening and/or a positive pregnancy test (serum and/or urine) on Day -1 in women of childbearing potential.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest.
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF [QTc corrected using Fridericia's formula] >450 ms, complete left bundle branch block (LBBB), signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third- degree AV (atrioventricular) block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with defined abnormalities in kidney and liver laboratory tests at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-04-17 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Mouth Feel Effect | 1, 5, 10, 20 minutes post dose
  Mouth feel visual analogue scale (VAS) assesses the participant's global perception of mouth feel (that is, effects over the whole course of the drug experience including any carryover effects). A 100-point VAS is used to assess response based on a score ranging from 0 points to 100 points (0 points = " Bad Mouth feel ", 50 points = "neither bad nor good mouth feel", and 100 points = "Good Mouth feel ").
Part 1: Bitter effect | 1, 5, 10, 20 minutes post dose
  Bitter visual analogue scale (VAS) assesses the participant's global perception of bitterness (that is, effects over the whole course of the drug experience including any carryover effects). A 100-point VAS is used to assess response based on a score ranging from 0 points to 100 points (0 points = " extremely bitter ", 50 points = "neither bad nor good bitterness", and 100 points = "not bitter").
Part 1: Tongue/mouth burn effect | 1, 5, 10, 20 minutes post dose
  Tongue/mouth burn visual analogue scale (VAS) assesses the participant's global perception of tongue/mouth burn (that is, effects over the whole course of the drug experience including any carryover effects). A 100-point VAS is used to assess response based on a score ranging from 0 points to 100 points (0 points = "extreme burn", 50 points = "neither bad nor good burn", and 100 points = "no burn").
Part 1:Overall liking effect | 1, 5, 10, 20 minutes post dose
  Overall liking visual analogue scale (VAS) assesses the participant's global perception of overall liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100-point VAS is used to assess response based on a score ranging from 0 points to 100 points (0 points = "bad", 50 points = "neither bad nor good", and 100 points = "good").
Part 2: Area under the Concentration-Time Curve (AUC 0-144) of osivelotor, as data permits | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  AUC from 0 to 144 hours is a measure of the whole blood concentration of the drug over time. It is used to characterize drug absorption; if AUC0-144 not available, then AUClast will be calculated.

SECONDARY OUTCOMES:
Part 1: Number of Participants With Treatment-Emergent Adverse Events (AEs) | Day 1 to 28
Part 2: Number of Participants With Treatment-Emergent Adverse Events (AEs) | Day 1 to 84
Part 1 and 2: Number of participants with clinically significant laboratory abnormalities. | Day 1 to Day 2 for Part 1, Day 1 to Day 7 for Part 2.
Part 1: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | Day 1 and Day 2
Part 2: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | Day 1 and Day 7
Part 1: Number of Participants With Clinically Significant With Clinically Significant Vital Signs | Day 1 and Day 2
Part 2: Number of Participants With Clinically Significant With Clinically Significant Vital Signs | Day 1, 2 and Day 7
Part 2: Maximum observed whole blood concentration (Cmax) of osivelotor pediatric formulation | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Cmax is a measure of the highest whole blood concentration of the drug over time.
Part 2: Area under the Concentration-Time Curve (AUC last) of osivelotor | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  AUC from 0 hours to last value is a measure of the whole blood concentration of the drug over time. It is used to characterize drug absorption.
Part 2: Time (Tmax) to maximum observed whole blood concentration (Cmax) of osivelotor pediatric formulation | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Tmax is a measure of the time it takes to get to the highest whole blood concentration of the drug over time.
Part 2: Maximum observed whole blood concentration (Cmax, dose normalized, if applicable) of osivelotor pediatric formulation | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  Cmax is a measure of the highest whole blood concentration of the drug over time.
Part 2: Area under the Concentration-Time Curve (AUC last, dose normalized, if applicable) of osivelotor | 0, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144 hours post-dose
  AUC from 0 hours to last value is a measure of the whole blood concentration of the drug over time. It is used to characterize drug absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5351009